CLINICAL TRIAL: NCT04422769
Title: Tracking Needs of Persons with a Spinal Cord Injury (SCI) During the COVID-19 Pandemic
Brief Title: Needs of Persons with Spinal Cord Injury (SCI)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Kerri Morgan, Assistant Professor of Occupational Therapy and Neurology, Washington University School of Medicine
Other Study IDs: 202005026
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Persons with spinal cord injury (PwSCI) are at a greater risk for major health conditions and poorer health outcomes than persons without spinal cord injury (SCI). They often experience a great deal of health needs both on a physiological level as well as a psychosocial level. PwSCI frequently require supports and services to be able to live independently within the community. These services and supports are sometimes difficult to access within the community when the country is operating under regular capacity, in current times with the global COVID-19 pandemic, the challenges for obtaining and accessing supports and services will become much greater. The proposed project aims to identify the specific needs during this time of crisis and to provide referrals and resources to ameliorate those needs by surveying PwSCI in the St. Louis region. The project also hopes to determine if these persons experience isolation during shelter at home orders. PwSCI, who the investigators serve or have served in the past, will be contacted via phone or e-mail once a month for six months and asked to complete a questionnaire that will allow the investigators to track the participant's needs during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Acquiring a spinal cord injury (SCI) can be a traumatic event resulting in significant life changes. Both the physical and psychosocial consequences of spinal cord injury may negatively impact one's ability to accomplish activities of daily living, fully participate in occupations, and fulfill social roles. People with SCI are at a greater risk for major health conditions such as heart disease, high blood pressure, obesity, and diabetes than the population without disabilities. Approximately 30% of individuals with SCI are also at risk for developing negative mood states that include depression, anxiety, and anger. These negative mood states can also increase the risk of poor health outcomes, including increased medical complications, decreased independence in self-care, and decreased productivity. People with SCI also often require a great deal of supports and services to live independently within the community, such as a personal care attendant to assist with activities of daily living, access to accessible transportation, access to medical care, and access to repair services for their mobility device. Many of these supports and services are difficult to obtain in the community, medical institutions, and businesses when everything is operating in a regular capacity. With the changes in daily operations related to the COVID-19 pandemic there are many concerns about whether vulnerable populations like persons with SCI will be able to access the supports and services they need, this project will give the investigators information about what the needs are and whether they are being met.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of an SCI; are 18 years or older; live in the community in the Greater St. Louis area, and have the ability to understand English.

Exclusion Criteria:

* cognitive impairment that does not allow them to provide consent and/or ability to understand the questions posed in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of two hundred and fifty (n=250) persons with SCI will be recruited from the St. Louis, MO community. Many of these persons will be those who have participated in some of the investigators other research projects in the past. We also have collaborations with the Washington University Seating and Mobility Clinic and Paraquad, the local center for independent living.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
NIH Toolbox Instrumental Support Survey - change in instrumental support | Baseline, 3 month and 6 month
  Instrumental Support refers to the perception that people in one's social network are available to provide material or functional aid in completing daily tasks (such as making meals or providing transportation) if needed. This self-report measure for adults (ages 18 and above) is an 8-item calibrated scale.This study will use the measure to determine if people's instrumental support changes during a pandemic.

SECONDARY OUTCOMES:
UCLA (University of California - Los Angeles) 3-item Loneliness Scale - change in social isolation | Baseline, 3 month and 6 month
  A scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each of the 3 items as hardly ever (score of "1"), some of the time (score of "2"), or often (score of "3"). The scores for each individual question can be added together to give you a possible range of scores from 3 to 9. The higher the score the more lonely the person will be. This study will use the measure to determine if people feel socially isolated during a pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri A Morgan, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Adnana Y, Mckenzie A, Miyahara M. Self-efficacy for quad rugby skills and activities of daily living. Adapted Physical Activity Quarterly. 2001; 18: 90-101.
- [Background] Blauwet C, Willick SE. The Paralympic Movement: using sports to promote health, disability rights, and social integration for athletes with disabilities. PM R. 2012 Nov;4(11):851-6. doi: 10.1016/j.pmrj.2012.08.015. PMID 23174549
- [Background] Slater D, Meade MA. Participation in recreation and sports for persons with spinal cord injury: review and recommendations. NeuroRehabilitation. 2004;19(2):121-9. PMID 15201471
- [Background] U.S. Department of Health and Human Services. (2000). Healthy people 2010: Understanding and improving health. 2nd ed. Washington, DC: U.S. Government Printing Office.
- [Background] Jacobs PL, Beekhuizen KS. (2005). Appraisal of physiological fitness in persons with spinal cord injury. Topics in Spinal Cord Injury Rehabilitation, 10(4):32-50.
- [Background] Keyser RE, Rasch EK, Finley M, Rodgers MM. Improved upper-body endurance following a 12-week home exercise program for manual wheelchair users. J Rehabil Res Dev. 2003 Nov-Dec;40(6):501-10. doi: 10.1682/jrrd.2003.11.0501. PMID 15077662
- [Background] Post MW, van Leeuwen CM. Psychosocial issues in spinal cord injury: a review. Spinal Cord. 2012 May;50(5):382-9. doi: 10.1038/sc.2011.182. Epub 2012 Jan 24. PMID 22270190
- [Background] Middleton J, Tran Y, Craig A. Relationship between quality of life and self-efficacy in persons with spinal cord injuries. Arch Phys Med Rehabil. 2007 Dec;88(12):1643-8. doi: 10.1016/j.apmr.2007.09.001. PMID 18047880